CLINICAL TRIAL: NCT04142359
Title: A Pharmacokinetic Sub-Study of QUILT-3.032 (CA ALT-803-01-16): A Multicenter Clinical Trial of Intravesical Bacillus Calmette-Guerin (BCG) in Combination With ALT-803 in Patients With BCG Unresponsive High Grade Non-Muscle Invasive Bladder Cancer and QUILT-2.005: A Study of Intravesical BCG in Combination With ALT-803 in Patients With Non-Muscle Invasive Bladder Cancer
Brief Title: PK Sub-Study of QUILT-3.032 (CA ALT-803-01-16) and of QUILT-2.005 (CA ALT-803-01-14)
Status: Terminated | Type: Observational
Why Stopped: Study was closed due to the recent pandemic and enrollment challenges.
Sponsor: Altor BioScience (Industry)
Responsible Party: Sponsor
Other Study IDs: QUILT-3.032-2.005-PK
Record Dates: First submitted 2019-10-23; First posted 2019-10-29 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2021-01

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — ALT-803

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: CIS (either study): Patients with histologically confirmed presence of BCG-unresponsive CIS, [with or without Ta/T1 papillary disease].
  Interventions: Biological: BCG in Combination with N-803
- Cohort B: High-Grade Ta/T1 Papillary Disease (either study): Patients with histologically confirmed presence of BCG-unresponsive high-grade Ta/T1 papillary disease
  Interventions: Biological: BCG in Combination with N-803
- Cohort C: CIS (QUILT-3.032): Patients with histologically confirmed presence of BCG-unresponsive CIS, [with or without Ta/T1 papillary disease].
  Interventions: Drug: N-803 alone

INTERVENTIONS:
Biological: BCG in Combination with N-803 — BCG in Combination with N-803
  Other Names: N-803
  Groups: Cohort A: CIS (either study); Cohort B: High-Grade Ta/T1 Papillary Disease (either study)
Drug: N-803 alone — N-803 alone
  Groups: Cohort C: CIS (QUILT-3.032)

SUMMARY:
Non-interventional PK sub-study of QUILT-3.032 (CA-ALT-803-01-16) and QUILT-2.005 (CA-ALT-803-01-14)

DETAILED DESCRIPTION:
QUILT-3.032 is a Phase 2, open-label, single-arm, three-cohort, multicenter study of intravesical BCG plus ALT-803 in patients with BCG unresponsive high grade NMIBC. Patients will be enrolled into one of three study cohorts. Cohort A will enroll 80 patients who have histologically confirmed presence of BCG-unresponsive carcinoma in situ (CIS) [with or without Ta or T1 disease]. Cohort B will enroll 80 patients who have histologically confirmed BCG-unresponsive high-grade Ta or T1 disease. Cohort C will enroll up to 23 patients who also have histologically confirmed presence of BCG-unresponsive CIS [with or without Ta/T1 papillary disease]. Patients in Cohorts A and B will receive ALT-803 plus BCG combination treatment. Patients in Cohort C will receive ALT-803 alone. Enrollment of Cohort C will start once the enrollment of Cohort A is complete. Cohorts A, B, and C are independent study cohorts and will be separately evaluated for efficacy. All patients treated in the study will receive via a urinary catheter in the bladder, BCG plus ALT-803 or ALT-803 alone weekly for 6 consecutive weeks during the induction treatment period.

QUILT-2.005 is a phase 2b, randomized, two-cohort, open-label, multicenter study of intravesical ALT-803 plus BCG versus BCG alone, in BCG naïve patients with high-grade NMIBC. Patients will be enrolled into one of two study cohorts and randomized into two arms to be treated with either ALT-803 plus BCG or BCG alone. Cohort A will initially enroll 366 patients who have histologically confirmed CIS (with or without Ta/T1 papillary disease). Cohort B will initially enroll 230 patients who have histologically confirmed high-grade papillary Ta/T1 disease only. Cohorts A and B are two independent study cohorts and will be evaluated separately for efficacy.

PK sub-study: Blood samples to determine serum levels of ALT-803 will be collected on study day 1 prior to dosing, and at post-bladder voiding (+ 15 minutes), 24 (±2), 48 (±4), 72 (±4), 96 (±4) and 168 (±4) hours after dosing administered at study Week 1 and again at the same time points for study Week 6. Six subjects from either cohort A (either study) or cohort C (QUILT 3.032) and six subjects from cohort B (either study) will be sampled initially. Up to an additional 4 subjects for each cohort may also be sampled. Patients enrolled in QUILT 2.005 must have been randomized to receive ALT-803 plus BCG to be eligible for the PK sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who are eligible for and have entered into protocol QUILT-3.032 or QUILT-2.005 may participate in this sub-study.
* Patients enrolled in QUILT-2.005 must have been randomized to receive ALT-803 plus BCG to participate in this sub-study.

Exclusion Criteria:

* Refusal to provide voluntary written informed consent and HIPAA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations.
* Loss of ≥ 475 mL blood volume or blood transfusion of any blood product within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six subjects from either Cohort A (either study) or Cohort C (QUILT-3.032) and six subjects from Cohort B (either study) will be sampled initially in this PK sub-study. Up to an additional 4 subjects from each cohort may also be sampled.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Garner, PhD, Study Director — ImmunityBio, Inc.
Locations (6):
- United States (6):
  - UCLA Department of Urology, Los Angeles, California
  - University of Miami Miller School of Medicine-Sylvester Comprehensive Cancer Center, Miami, Florida
  - Adult & Pediatric Urology, Omaha, Nebraska
  - NYU Winthrop University Hospital Department of Urology, Garden City, New York
  - Manhattan Medical Research, New York, New York
  - Virginia Urology, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8096327/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032) | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (NA) — Only 1 participant was enrolled in the study. |  |  | 73 (NA) — Only 1 participant was enrolled in the study.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Non-muscle invasive bladder cancer enrolled on either QUILT-3.032 or QUILT-2.005 [Count of Participants; unit: Participants] | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Half-life (t½)
Description: Half-life (t½)
Time Frame: Study day 1 prior to dosing, and at post-bladder voiding (+ 15 minutes), 24 (±2), 48 (±4), 72 (±4), 96 (±4) and 168 (±4) hours after dosing administered at study Week 1 and again at the same time points for study Week 6.
Population: Systemic N-803 was below the limit of quantitation for all subjects at all time points assessed. Following intravesical administration, there was no evidence of systemic N-803 in any subject. PK parameters were not calculated.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
Hours | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

2. Primary Outcome: Apparent (Extravascular) Volume of Distribution (Vz/F)
Description: Apparent (extravascular) volume of distribution (Vz/F)
Time Frame: Study day 1 prior to dosing, and at post-bladder voiding (+15 minutes), 24 (±2), 48 (±4), 72 (±4), 96 (±4) and 168 (±4) hours after dosing administered at study Week 1 and again at the same time points for study Week 6.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
mL/kg | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

3. Primary Outcome: Apparent (Extravascular) Clearance (CL/F)
Description: Apparent (extravascular) clearance (CL/F)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/day/kg
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
L/day/kg | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

4. Primary Outcome: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
pg/mL | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

5. Primary Outcome: Time of the Observed Maximum Concentration (Tmax)
Description: Time of the observed maximum concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
Days | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

6. Primary Outcome: Area Under the Plasma Concentration Curve From Time 0 Through the Last Measurable Concentration (AUC0-t)
Description: Area under the plasma concentration curve from time 0 through the last measurable concentration (AUC0-t)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Day*pg/mL
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
Day*pg/mL | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

7. Primary Outcome: Area Under the Plasma Concentration Curve From Time 0 Extrapolated to Infinite Time (AUC0-inf)
Description: Area under the plasma concentration curve from time 0 extrapolated to infinite time (AUC0-inf)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Day*pg/mL
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
Number analyzed (Participants) | 1 | 0 | 0
Day*pg/mL | NA (NA) — Systemic N-803 was below the limit of quantitation at all time points assessed. Thus, there was no evidence of systemic N-803 exposure after intravesical administration. |  |

ADVERSE EVENTS:
Description: Any AEs that occurred during the sub-study and were associated with QUILT-3.032 were to be collected and handled per the QUILT-3.032 protocol. This PK sub-study was designed to evaluate the pharmacokinetic (PK) profile of intravesical N-803 in combination with BCG in patients with high grade NMIBC. All AEs were to be reported in the respective main studies, and the only data collected in this study were related to the primary endpoints in QUILT-3.032-2.005-PK.
Arm/Group | Cohort A: CIS (Either Study) | Cohort B: High-Grade Ta/T1 Papillary Disease (Either Study) | Cohort C: CIS (QUILT-3.032)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT04142359/Prot_SAP_000.pdf